CLINICAL TRIAL: NCT04004442
Title: Phase I Study of Avelumab in Combination With AXL Inhibitor AVB-S6-500 in Patients With Advanced Urothelial Carcinoma
Brief Title: Avelumab in Combination With AVB-S6-500 in Patients With Advanced Urothelial Carcinoma
Acronym: COAXIN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Aravive, Inc. (Industry); EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-COAXIN
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma
Keywords: avelumab; AVB-S6-500; renal pelvis cancer; ureter cancer; urinary bladder cancer; urethra cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Ureteral Neoplasms; Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab + AVB-S6-500 (Experimental)
  Interventions: Drug: Avelumab; Drug: AVB-S6-500

INTERVENTIONS:
Drug: Avelumab — Avelumab: 800 mg IV every two weeks (on days 1 and 15 of a 28-day cycle)
Drug: AVB-S6-500 — AVB-S6-500: 10mg/kg IV every 2 weeks (on days 1 and 15 of a 28-day cycle) Potential dose reduction: AVB-S6-500: 5mg/kg IV weekly (on days 1, 8, 15 and 22 of a 28-day cycle)

SUMMARY:
The purpose of this research study is to test the safety of avelumab and AVB-S6-500 and see what effects (good and bad) this combination treatment has on patients with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
Patients will have tests and exams to see if they are eligible for the clinical trial. If found eligible, the patient will receive treatment with avelumab and AVB-S6-500 by vein once every two weeks.

This study has two parts in order to determine the maximum tolerated dose of AVB-S6-500. If the patient is enrolled on the first dose level, the patient will be treated at a higher dose every two weeks with AVB-S6-500. If the patient is enrolled on the second dose level, the patient will be receive AVB-S6-500 only once a week at a lower dose. The patient would continue to receive avelumab twice weekly at the same dose.

Patients will receive the study treatment as long as there is evidence that the tumor is not growing or spreading and they are not having any unacceptable, bad side effects.

Patients will be monitored during treatment with tests and exams and after treatment completion for up to one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histologically confirmed locally advanced unresectable (T4b or N2/N3 disease) or metastatic urothelial cancer (including renal pelvis, ureters, urinary bladder, urethra).
3. Eligible patients must have had either:

   1. Progressed after treatment with at least 1 prior platinum-containing regimen, (e.g., received at least 2 cycles of cisplatin or carboplatin-based regimen) for inoperable locally advanced unresectable or metastatic urothelial carcinoma, OR OR
   2. Experienced disease progression or recurrence within 12 months of completion of neoadjuvant or adjuvant cisplatin-based chemotherapy, OR OR
   3. Ineligible for cisplatin-based chemotherapy due to eastern co-operative oncology group (ECOG) performance status 2, grade ≥2 neuropathy, GFR<60 mL/min, grade ≥2 hearing loss or New York Heart Association class III or worse congestive heart failure.
   4. Declined platinum (cisplatin or carboplatin) based chemotherapy after informed discussion with the treating investigator
4. Available pretreatment baseline tumor specimen or willingness to undergo biopsy of primary or metastatic lesion if archived specimen is not available.
5. ECOG performance status of ≤2
6. At least one measurable lesion by RECIST version 1.1
7. Patients who are able to understand and sign the informed consent form.
8. Ability to comply with protocol
9. Adequate hematologic and end-organ function per protocol
10. For women of childbearing potential: Negative serum or urine pregnancy test at screening.
11. For both male and female subjects: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 30 days after the last dose of study drug

Exclusion Criteria:

1. Concurrent systemic treatment with an anticancer treatment or investigational drug within 28 days. Palliative radiation to symptomatic primary tumor or metastases is permitted as long as there are other measurable lesions present outside of the radiation field.
2. Prior therapy with anti-PD-1 or PD-L1 agents.
3. Concurrent systemic therapy with corticosteroids (>10 mg prednisone equivalent) or other immunosuppressive agents within 28 days before starting trial drug. Short-term administration of systemic steroids (less than 7 days), adrenal replacement steroid doses (≤10 mg daily prednisone equivalent), topical, intranasal and inhaled steroid use is permitted.
4. Patients with untreated or symptomatic central nervous metastases will be excluded. Patients appropriately treated with either surgery and/or radiation therapy will be eligible to participate in the study 4 weeks after completion of radiation/surgery and if follow up brain imaging after CNS directed therapy demonstrates stability or improvement in brain metastases.
5. Active second malignancy or previous history of malignant disease (other than urothelial carcinoma) diagnosed within the last 3 years, with the exclusion of basal or squamous cell carcinoma of the skin, cervical carcinoma in situ and pT2 prostate adenocarcinoma with Gleason score ≤7 (with no dominant pattern 4).
6. Prior organ transplantation, including allogenic stem-cell transplantation.
7. Known history of HBV infection (including acute and chronic infection) and untreated hepatitis C. Patients with treated HCV infection will be eligible.
8. Known hypersensitivity to monoclonal antibody or any biologic drug, history of anaphylaxis, or uncontrolled asthma.
9. Persisting toxicity related to prior therapy that was > grade 1 according to NCI-CTCAE v4; grade ≤2 sensory neuropathy is allowed.
10. Pregnant or lactating, or intending to become pregnant during the study

    a. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative pregnancy test result within 14 days prior to the first dose of study treatment.
11. Diagnosis of active autoimmune disease requiring systemic immunosuppression. Patients with type 1 diabetes, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring systemic immunosuppression are eligible.
12. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

    a. History of radiation fibrosis in the radiation field (fibrosis) is permitted.
13. Active infection requiring systemic therapy.
14. Severe infections within 4 weeks prior to the first dose of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
15. Administration of a live/attenuated vaccine within 4 weeks prior to the first dose of study treatment, within 5 months following the administration of the last dose of study drug, or anticipation that such a live/attenuated vaccine will be required during the study.
16. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | up to 2 years
  To investigate the safety and tolerability of the study drug combination for Avelumab with AVB-S6-500

SECONDARY OUTCOMES:
Progression Free Survival | up to two years
  period from the time of patient enrollment until disease progression, death, or date of last contact or to the date of censoring (dropout, end of study or death)
Clinical Benefit Rate | up to two years
  proportion of patients with complete or partial response, or stable disease per RECIST 1.1 on treatment with avelumab and ABV-S6-500
Duration of Response | up to two years
  defined as the period from the date of confirmed tumor response until disease progression, death, or date of last contact or to the date of censoring (dropout, end of study or death)
Overall Survival | up to two years
  the period from patient enrollment until death, or date of last contact or to the date of censoring (end of study)
Investigator assessed Objective Response Rate | up to 2 years
  To evaluate the antitumor efficacy of avelumab and AVB-S6-500 as measured by the objective response rate assessed by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Tripathi, MD, Principal Investigator — Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No